CLINICAL TRIAL: NCT01382459
Title: The Efficacy of Constructed Intervention by Home and School Visits by Diabetes Nurses on Diabetic Control of Children With Type I Diabetes
Brief Title: Constructed Intervention by Home and School Diabetes Nurse Visits on Diabetic Control of Children With Type I Diabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Collaborators: Clalit Health Services (Other)
Responsible Party: Prof. Eli Hershkovitz, Pediatric endocrinology and diabetes unit
Other Study IDs: sor517111ctil
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: children
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- type 1 DM children- intervention group: will have home visits and trainings at school
- type 1 DM children- control group: will receive the standard care at the clinic

SUMMARY:
The investigators assume that an intervention program that includes home visits and trainings of diabetes' nurse and dietitian will lead to an improvement of the patients' metabolic balance, a decrease in complications' rate, a reduction of hospitalizations and an economic streamlining.

DETAILED DESCRIPTION:
The investigators assume that during the study, subjects from the intervention group will reach a better metabolic balance than the control group. In this group the following changes will occur:

* A decrease in HbA1C levels.
* A decrease in Hypoglycemia events.
* A decrease in DKA events.
* A decrease in patients' visits in ER and hospitalizations.
* An improvement in the knowledge of the patients and their families about the disease.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 DM diagnosis from at least 8 months/
* HbA1C levels >8
* Signed inform consent.

Exclusion Criteria:

- Children who are not in educational settings and are not hebrew or arabic speakers.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: type 1 DM children in the age of 4-18, living in Beer Sheva and the area, who are under treatment in the pediatric diabetes unit in Soroka.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-07

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka medical center, Beersheba, Israel, Israel